CLINICAL TRIAL: NCT05218772
Title: Objective and Perceived Health Status of Elderly People With Moderate or Severe Haemophilia in France: an Ancillary Study of the FranceCoag Registry
Acronym: SENIORHEMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-20
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Moderate or Serious Haemophilia
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly people with moderate or severe haemophilia
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Each eligible participant will receive a questionnaire to complete concerning: objective health status; perceived health status (QoL assessed by the WHOQOL-Old questionnaire); demographic data; social data; psycho-cognitive data (anxious symptoms, depressive symptoms, use of coping strategies, time perspective)

SUMMARY:
Background:

Elderly people with serious haemophilia (PwSH), i.e., with moderate or severe haemophilia, have major comorbidities due to consequences of haemophilia. Also, the comorbidities related to age are added. Despite the existence of numerous studies on the objective health status of elderly PwSH, some limitations may be stated (need to update the results in a more contemporary context, no studies conducted in France, highlighted determinants focused on demographic and clinical factors).

On the contrary, the perceived health status of elderly PwSH has been little described. Only two studies specifically addressed the quality of life (QoL) of elderly PwSH. These studies reported an altered QoL in some domains, in comparison with reference values from the general population. However, some limitations may also be stated (need to bring results in a more contemporary context, no studies conducted in France, highlighted determinants focused on clinical factors).

Since serious haemophilia is a rare disease, studies are often performed on a small number of subjects. The present project relies on the FranceCoag registry, a unique exhaustive national cohort of PwSH followed over time among whom 612 are elderly PwSH.

Objectives:

Main objective: to describe the objective and perceived health status of elderly (≥60 y.o.) PwSH from of a French exhaustive national registry, and to compare their health status with that of the French general elderly population.

Secondary objective: to identify individual (demographic, clinical, social, psycho-cognitive) and collective characteristics (related to healthcare organisation), associated with the objective and perceived health status of elderly PwSH in France.

Materials and Methods:

A national, multicentric, observational, cross-sectional study will be conducted. It will be based on the participation of elderly PwSH already included in the FranceCoag registry. Each eligible participant will receive a questionnaire to complete concerning: objective health status; perceived health status (QoL assessed by the WHOQOL-Old questionnaire); demographic data; social data; psycho-cognitive data (anxious symptoms, depressive symptoms, use of coping strategies, time perspective). Therapeutic and clinical data related to haemophilia will be collected via the FranceCoag registry database. Data concerning healthcare organisation will be collected directly from investigators of Haemophilia Treatment Centres.

The main analysis will consist in the description and comparison of the health status with reference data from the French general elderly population. Standardisation methods will be used to take into account a potential imbalance between the study population and the reference population, related to age and especially to sex, as haemophilia is a predominantly male disease.

The secondary analysis will consist in the identification of potential determinants of the health status. Structural equation models will be performed to take into account the complexity of the relationships between the determinants.

Impact of the proposal Better understanding the impact of the disease on patients' experience is essential in a systematic global perspective of health, that aims to care and support the individual not only as a patient but also as a person in his/her environment. This study based on a registry will allow to improve the knowledge by updating literature data on the health status of elderly PwSH, adding elements to the rare literature data on the perceived health status, providing data in the French specific context, and identifying both classical and more original determinants of health status of elderly PwSH. These results will be used to better identify elderly PwSH at high risk of poor health status, to propose recommendations and to set up actions to offer them an adapted support, and to elaborate new versions of public health plans dedicated to haemophilia or to rare diseases.

ELIGIBILITY:
Inclusion Criteria:

* People with serious haemophilia, i.e., with (A or B) moderate or severe haemophilia;
* People aged 60 years or over;
* People included in the FranceCoag registry;
* People followed in one of the Haemophilia Treatment Centre participating in the study;
* People who do not oppose to participate in the study.

Exclusion Criteria:

* People with comprehension disabilities;
* Participants who a posteriori oppose to participate in the study.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly people with moderate or severe haemophilia in France
Sampling Method: Non-Probability Sample
Enrollment: 612 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective health status (apart from serious haemophilia) | 1 day
  Declaration by the participant of at least one chronic disease or health issue (apart from serious haemophilia)
Perceived health status | 1 day
  Assessed by the quality of life, which will be measured by the WHOQOL-Old questionnaire

CONTACTS AND LOCATIONS:
Locations (28):
- France (28):
  - Chu Amiens, Amiens
  - Ch Annecy - St Julien, Annecy
  - Chu de Besancon, Besançon
  - Chu de Bordeaux, Bordeaux
  - Chu Brest, Brest
  - Chu de Caen, Caen
  - Centre hospitalier Métropole Savoie, Chambéry
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu de Dijon, Dijon
  - Chu La Reunion, La Réunion
  - Chu Le Mans, Le Mans
  - Chru de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Ap-Hm, Marseille
  - Chu Montpellier, Montpellier
  - Chu de Nancy, Nancy
  - Chu Nantes, Nantes
  - Chu de Nice, Nice
  - AP-HP, Paris
  - Chu Poitiers, Poitiers
  - Chu Reims, Reims
  - Chu de Rennes, Rennes
  - Chu de Rouen, Rouen
  - Chu St Etienne, Saint-Etienne
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - Chru de Tours, Tours
  - Ch Versailles, Versailles